CLINICAL TRIAL: NCT04398030
Title: Randomized Crossover Euglycemic Clamp Study in Adult Patients With T1DM to Assess Pharmacokinetics and Pharmacodynamics of Subcutaneously Infused Insulin Using an Investigational Extended Wear Continuous Subcutaneous Insulin Infusion Cannula Compared to a Commercial Infusion Set
Brief Title: Pharmacokinetics (PK)/ Pharmacodynamics (PD) of an Extended Wear Infusion Set for Continuous Subcutaneous Insulin Infusion (CSII) in Type 1 Diabetes Mellitus (T1DM) Patients ("PEXIS")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capillary Biomedical, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); AMCR Institute (Other); Integrated Medical Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 150-1022-00; 2R44DK110969-02 (NIH)
Record Dates: First submitted 2020-05-08; First posted 2020-05-21 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- coil-reinforced soft polymer indwelling cannula (Experimental): Participants in this arm are randomized into the coil-reinforced soft polymer indwelling cannula group and then switched to a soft Teflon indwelling cannula group after a 2-week washout/rest (±1 week). The participant will try to wear each infusion set for 7 consecutive days.
  Interventions: Device: coil-reinforced soft polymer indwelling cannula
- soft Teflon indwelling cannula (Active Comparator): Participants in this arm are randomized into the soft Teflon indwelling cannula group and then switched to the coil-reinforced soft polymer indwelling cannula group after a 2-week washout/rest (±1 week). The participant will try to wear each infusion set for 7 consecutive days.
  Interventions: Device: soft Teflon indwelling catheter

INTERVENTIONS:
Device: coil-reinforced soft polymer indwelling cannula — Insulin infusion set will be used for up to 7 days of continuous use or until failure
  Arms: coil-reinforced soft polymer indwelling cannula
Device: soft Teflon indwelling catheter — Insulin infusion set will be used for up to 7 days of continuous use or until failure
  Arms: soft Teflon indwelling cannula

SUMMARY:
This study has been designed as a prospectively enrolled, randomized sequence, 2-way crossover study of device performance, tolerability and safety of an investigational insulin infusion set using a coil-reinforced soft polymer indwelling cannula versus a commercial insulin infusion set using a soft Teflon indwelling cannula, during two 7-day home use periods with 4 in-clinic euglycemic clamp sessions during each of the 7-day periods. After a wash-out period, subjects will cross over into the investigational or control group, respectively.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Participants are 18 - 70 years of age inclusive
2. Participant is in generally good health, as determined by the investigator
3. Participant is willing and able to individually complete written informed consent and agrees to comply with all study related testing and examinations
4. Participant must be geographically stable (e.g., expects to be available and capable of returning for all study specified test and examinations) during the study period
5. Participant has been diagnosed with T1DM for at least 12 months
6. C-peptide <0.6 nmol/L at screening
7. Participant has been using insulin pump therapy for at least 6 months and is currently using a Medtronic MiniMed pump, model series 530 or higher. Use of 670G in auto mode is acceptable.
8. Participant can provide a minimum of 14 days of insulin pump data to demonstrate pump use compliance
9. Participant is willing to perform frequent (4 times per day or more) self-monitoring of blood glucose (SMBG), including before meals and before bed, and using a meter and test strips provided by the sponsor during the two weeks of active treatment. This includes participants who are currently using real-time continuous glucose monitoring and may continue to do so, but must also collect SMBG values as instructed.
10. Participant is willing to perform serum ketone measurements whenever the blood glucose is determined to be greater than 250 mg/dL after extended fasting (e.g. overnight or more than five hours after a meal) using a ketone meter and strips provided by the sponsor
11. Participant has BMI in the range 20 - 35 kg/m2 inclusive
12. Participant has experience infusing a rapid-acting insulin analog for at least 6 months
13. Participant has been using or is willing to use a Continuous Glucose Monitor (CGM) (reading data available for at least 80% of time for a week of data collection during the screening period). Participants already using - Dexcom G6 real time CGM may continue to use their own CGM unit; participants not using the G6 will be provided with a G6 monitor. All participants will be provided with CGM disposables for use during the treatment period.
14. Participant has ability to understand and comply with protocol procedures and to provide informed consent
15. HbA1c ≤8.5%
16. Stable body weight in the 3 months prior to enrollment (change in body weight <5%)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Participants whose average total daily insulin dose exceeds 85 units/day (i.e., typically change insulin reservoirs more often than every 4 days on average)
2. Participants who routinely change their commercial insulin infusion sets on average less often than every 4.5 days
3. Female participant is pregnant or nursing
4. Participant has abnormal skin at intended device infusion sites (existing infection, inflammation, burns, or other extensive scarring)
5. Participant has hemoglobin <12.0 g/dL or potassium < 3.5 milliequivalent/L at screening
6. Participant has documented history in last 6 months of severe hypoglycemia associated with cognitive dysfunction sufficiently severe to require third party intervention or a history of impaired awareness of hypoglycemia.
7. Participant has a history of diabetic ketoacidosis in the last 6 months
8. Participant has known cardiovascular disease considered to be clinically relevant by the investigator
9. Participant has known arrhythmias considered to be clinically relevant by the investigator
10. Participant has known history of:

    1. Cushing's Disease,
    2. Pancreatic islet cell tumor, or
    3. Insulinoma
11. Participant has:

    1. Lipodystrophy,
    2. Extensive lipohypertrophy, as assessed by the investigator
12. Participant is undergoing current treatment with:

    1. Systemic oral or intravenous corticosteroids,
    2. Monoamine oxidase (MAO) inhibitors,
    3. Non-selective systemic beta-blockers,
    4. Growth hormone,
    5. Thyroid hormones, unless use has been stable during the past 3 months
    6. SGLT2 inhibitors
13. Participant has significant history of any of the following, that in the opinion of the investigator would compromise the participant's safety or successful study participation:

    1. Alcoholism,
    2. Drug abuse
14. Significant acute or chronic illness, that in the investigator's opinion, might interfere with participant safety or integrity of study results
15. Planned operation, MRI or CT which require removal of infusion set or CGM sensor during wear periods
16. Current treatment with systemic (oral or IV) corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, growth hormone, herbal products that, in the opinion of the investigator, may alter insulin sensitivity or confer undue risk to the participant's participation in the study or non-routine vitamins. Furthermore, thyroid hormones are not allowed unless the use of these has been stable during the past 3 months.
17. Current participation in another clinical drug or device study
18. Inability of the participant to comply with all study procedures or to understand the participant instructions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kastner JR, Bailey TS, Strange P, Shi L, Oberg KA, Strasma PJ, Joseph JI, Muchmore DB. Progressive Acceleration of Insulin Exposure Over 7 Days of Infusion Set Wear. Diabetes Technol Ther. 2023 Feb;25(2):143-147. doi: 10.1089/dia.2022.0323. Epub 2022 Dec 20. PMID 36342853
- See also: Site link which allows for the participant to enter information for the site to identify possible studies for participant enrollment — http://myamcr.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from the existing Type 1 diabetes database at the study center and from referrals from other diabetes treatment clinics in surrounding areas.
Groups:
- Coil-Reinforced Soft Polymer Indwelling Cannula Then Soft Teflon Indwelling Cannula: Participants in this arm are randomized into the coil-reinforced soft polymer indwelling cannula group and then switched to a soft Teflon indwelling cannula group after a 2-week washout/rest (±1 week). The participant will try to wear each infusion set for 7 consecutive days.
  Coil-reinforced soft polymer indwelling cannula: Insulin infusion set will be used for up to 7 days of continuous use or until failure
- Soft Teflon Indwelling Cannula Then Coil-Reinforced Soft Polymer Indwelling Cannula: Participants in this arm are randomized into the soft Teflon indwelling cannula group and then switched to the coil-reinforced soft polymer indwelling cannula group after a 2-week washout/rest (±1 week). The participant will try to wear each infusion set for 7 consecutive days.
  Soft Teflon indwelling catheter: Insulin infusion set will be used for up to 7 days of continuous use or until failure
Period: Treatment Period 1 (1 Week)
Arm/Group | Coil-Reinforced Soft Polymer Indwelling Cannula Then Soft Teflon Indwelling Cannula | Soft Teflon Indwelling Cannula Then Coil-Reinforced Soft Polymer Indwelling Cannula
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Coil-Reinforced Soft Polymer Indwelling Cannula Then Soft Teflon Indwelling Cannula | Soft Teflon Indwelling Cannula Then Coil-Reinforced Soft Polymer Indwelling Cannula
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Treatment Period 2 (1 Week)
Arm/Group | Coil-Reinforced Soft Polymer Indwelling Cannula Then Soft Teflon Indwelling Cannula | Soft Teflon Indwelling Cannula Then Coil-Reinforced Soft Polymer Indwelling Cannula
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to either the soft Teflon indwelling cannula group or the coil-reinforced soft polymer indwelling cannula group in treatment period 1. Then after a 2-week washout/rest (±1 week), participants crossed over into treatment period 2 using either the soft Teflon indwelling cannula or the coil-reinforced soft polymer indwelling cannula. The participant wore each infusion set up to 7 consecutive days in each treatment period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.6 (3.81)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Rate of Decline (s) Over Wear Time (DOI, Day 3, Day 5, Day 7) of the Natural Logarithm of the Area Under the Glucose Infusion Rate Curve [ln (AUC0-300(GIR))].
Description: The primary endpoint will be compared between the treatment groups.
Time Frame: 7 days
Population: Intent to Treat (ITT) population
Measure: Mean (95% Confidence Interval); unit: Slope
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
Slope | -0.102 [-0.220 to 0.016] | -0.097 [-0.213 to 0.019]

2. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Time-to-Maximum Insulin Concentration (Tmax)
Description: The Time-to-Maximum Glucose Infusion (GIR) rate, tmax (GIR) is the minute between the time corresponding to the GIR max and Time 0.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
min
  Day 0 | 65.8 (30.07) | 67.5 (25.05)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 25.0 (7.07) | 31.0 (16.73)

3. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Maximum Insulin Concentration (Cmax)
Description: Cmax is the maximum insulin concentration between t=0 (bolus) and t=300 minutes.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
mU/L
  Day 0 | 57.8 (21.51) | 62.3 (20.94)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 86.6 (23.95) | 96.9 (49.12)

4. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Time-to-50% (Early) Maximum Insulin Concentration [t50%(Early)]
Description: The time to half-maximal insulin concentration- early (before peak)
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
min
  Day 0 | 22.8 (11.34) | 29.1 (10.59)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 11.5 (4.13) | 14.8 (5.21)

5. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Mean-residence Time (MRT) of Insulin
Description: Mean residence time quantifies the sum of average absorption time and average systemic residence time.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
min
  Day 0 | 121.8 (25.10) | 117.7 (27.08)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 77.4 (8.92) | 75.9 (14.07)

6. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Area Under the Curve (AUC0-300)
Description: The area under the insulin concentration curve until 300 minutes after bolus administration
Time Frame: 7 days
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mU*min/L
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
mU*min/L
  Day 0 | 9084 (2826) | 8982 (1453)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 6920 (1908) | 7313 (2483)

7. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Insulin Early Exposure: AUC0-60
Description: Area under the insulin concentration curve in the first 60 minutes after bolus administration
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: mU*min/L
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
mU*min/L
  Day 0 | 2131 (923.1) | 2200 (940.6)
  Day 7 | 3626 (922.9) | 3840 (2055)

8. Secondary Outcome: Mean Differences (Within Treatments Over Time Between Day 0 and Day 7) in Time-to-50% (Late) Maximum Insulin Concentration [t50%(Late)]
Description: Time at which 50% of the maximum insulin concentration was reached.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
Number analyzed (Participants) | 6 | 6
min
  Day 0 | 156.8 (34.13) | 156.5 (44.47)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 67.8 (13.20) | 76.3 (28.87)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Coil-reinforced Soft Polymer Indwelling Cannula | Soft Teflon Indwelling Cannula
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/6 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coil-reinforced Soft Polymer Indwelling Cannula (N=6) | Soft Teflon Indwelling Cannula (N=7)
Infusion Site Erythema (General disorders) | 1 (1) | 1 (1)
Infusion Site Induration (General disorders) | 1 (1) | 0 (0)
Infusion Site Edema (General disorders) | 1 (1) | 1 (1)
Infusion Site Pain (General disorders) | 1 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Participant-Device Interaction Incompatibility (Product Issues) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04398030/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04398030/SAP_001.pdf